CLINICAL TRIAL: NCT05115240
Title: The Effects of a Brief Mindfulness Intervention on Emotional Responses and the Moderating Role of Interoception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Mindfulness and interoception
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Whole Body Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Audio-guided mindfulness-based intervention (body scan) (Experimental)
  Interventions: Behavioral: Body Scan
- Enhanced Audio-guided mindfulness-based intervention (body scan) (Experimental): Participants undergo the same audio-guided body scan intervention. However, in this arm the instruction focuses on the positive effects of mindfulness-based interventions and body scan aiming to optimize participants' interventions outcome expectations of the intervention. The idea of this arm is to assess whether the effects of the mindfulness-based intervention can be augmented by boosting participants positive expectations prior to the intervention.
  Interventions: Behavioral: Body Scan
- Audio-Book (Active Comparator): Participants in this group listen to an audio-book for the same duration as the participants in the two experimental groups.
  Interventions: Other: Audio-book

INTERVENTIONS:
Behavioral: Body Scan — The body scan intervention aims to raise one's awareness of one's own body. It is considered a relaxation, meditation or mindfulness intervention. During the body scan participants will walk through his or her body by focusing their mind on specific body parts without analyzing, judging or reacting.
  Arms: Audio-guided mindfulness-based intervention (body scan); Enhanced Audio-guided mindfulness-based intervention (body scan)
Other: Audio-book — Participants listen to an audio book for the same amount of time as the body scan groups
  Arms: Audio-Book

SUMMARY:
This study examines the effects of a brief mindfulness intervention (body scan) on emotional responses (e.g., affect, heart rate variability (HRV)) compared to an active control group. Another aim is to assess whether the effects of the mindfulness intervention can be augmented by optimizing positive expectations. The moderating role of interception on the mindfulness intervention's effects will also be examined.

DETAILED DESCRIPTION:
This 3-armed study examines the effects of a brief mindfulness intervention (audio-guided body scan) on emotional responses (e.g., affect, and heart rate variability (HRV)) compared to an active control group (listening to an audio-book). Another aim is to assess whether the effects of the mindfulness intervention can be augmented by optimizing positive expectations. The moderating role of interception (i.e., interoceptive accuracy as assessed by the Schandry task) on the mindfulness intervention's effects will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* fluent in the German language
* ability to give informed consent

Exclusion Criteria:

* cardiovascular disease (previous myocardial infarction, hypertension)
* neurological disorders (epilepsy, stroke, multiple sclerosis)
* continuous medication intake (exceptions: contraceptives, nutritional supplements, L-thyroxine for hypothyroidism are allowed)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in affect | Change from pre (baseline) to post scores (30 minutes later)
  Participants are asked to rate adjectives regarding their current mood (positive and negative) at two time points (baseline and after body scan or active control intervention) on a questionnaire. Change scores are calculated (post- minus pre-scores).
  Instrument: Positive and Negative Affect Scale (PANAS) by Watson, Clark, and Tellegen (1988) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much). Range for sum score of positive/negative affect: 10-50. For positive affect higher scores are better; for negative affect lower scores are better.

SECONDARY OUTCOMES:
Change in perceived stress | Change from pre (baseline) to post scores (30 minutes later)
  Participants are asked to rate how stressed they feel at the moment at two time points (baseline and after body scan or active control intervention) on a questionnaire (VAS: item ranges from 0 (not stressed at all) - 100 (very stressed). Change scores are calculated (post- minus pre-scores). More negative change scores are better since it indicates a stronger stress reduction (maximum reduction: -100). Higher positive change scores are worse since this indicates an increase in perceived stress (maximum increase: +100). Range of change scores: -100 - +100).
Change in heart rate variability (HRV) | Change from pre (baseline) to post scores (30 minutes later)
  Heart rate variability (HRV) describes the variations between two successive heart beats and is considered a measure for cardiac adaptation to internal and external stimuli. HRV is considered an important transdiagnostic biomarker of health. HRV is frequently quantified using time- domain measures such as the standard deviation of NN intervals (SDNN) and the root mean square of successive differences between normal heartbeats (RMSSD). For HRV levels higher scores are better
Change in interoceptive accuracy | Change from pre (baseline) to post scores (30 minutes later)
  The heartbeat perception task (Schandry, 1981) encompasses several trials in which participants are instructed to silently count their heartbeats and report the number they counted after each trial. Reported and actual number of heart beats (as assessed by ECG) will be used to calculate a heartbeat detection index (error score).
Change in state anxiety and depression | Change from pre (baseline) to post scores (30 minutes later)
  The State-Trait-Anxiety-Depression-Inventory (STADI) (Laux, L. Hock, M., Bergner-Köther, R., Hodapp, V. & Renner, K., 2013) measures participants' state anxiety (10 items) and state depression (10 items) severity. Each item can be answered on a 4-point-scale from 1 (not at all) - 4 (very much). Sum scores are calculated and range from 10-40 for each scale (depression and anxiety). Lower scores indicate lower severity (i.e., less negative mood).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data will be shared with researchers providing a relevant and methodologically sound proposal